CLINICAL TRIAL: NCT03154268
Title: Retrospective Longitudinal Study of Gestational Weight Gain Among Chinese Pregnant Women
Acronym: GWGCPW
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Collaborators: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Jing Tan, Chinese Evidence-based Medicine Center, West China Hospital
Other Study IDs: GWG-China-2016
Record Dates: First submitted 2017-03-24; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Gestational Weight Gain
Keywords: Gestational weight gain; Chinese pregnant women; Retrospective longitudinal study; China; IOM guideline; Adverse outcome; Model
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the reference ranges and rates of gestational weight gain among Chinese pregnant women, and to analyze the correlation between gestational weight gain and adverse outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Deliveries between January 2013 and December 2014;
2. Gestational age between 37 weeks or older and less than 42 weeks;
3. Registration with care documents at the first prenatal visit prior to the 15th gestational week;
4. Had at least five follow-up visits until delivery.

Exclusion Criteria: None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese pregnant women who had deliveries at West China Women and Children's Hospital, Sichuan University
Sampling Method: Non-Probability Sample
Enrollment: 10422 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Preeclampsia | After 20th gestational weeks till delivery, about 5 months
  Maternal systolic pressure ≥140 mmHg and/or diastolic pressure ≥90 mmHg during gestation. Urine protein ≥5.0 g within 24h, urine volume <400 mL. HELLP syndrome or pulmonary edema present.
Eclampsia | After 20th gestational weeks till delivery, about 5 months
  Tonic-clonic seizures (convulsions) in preeclampsia patients, including convulsions and coma, not due to pre-existing or organic brain disorders.
ICP | After 14th gestational weeks till delivery, about 6 months
  Intrahepatic cholestasis of pregnancy.
Placenta previa | During pregnancy till delivery
  Placenta partially or entirely covered the lower uterine segment diagnosed using antenatal ultrasound.
Gestational diabetes | After 24th gestational weeks, about 4 months
  By oral glucose tolerance test between 24th and 28th gestational weeks (fasting glucose ≥5.1 mmol/L, 1-h glucose ≥10.0 mmol/L, 2-h glucose ≥8.5 mmol/L; one abnormal result sufficient).
Ruptured uterus | During delivery
  Rupture of maternal uterus confirmed by laparotomy.
Placental abruption | After 20th gestational weeks till delivery, about 5 months
  Abruption of a normally positioned placenta before delivery, diagnosed by clinical symptoms, ultrasound, fetal heart monitoring, or laboratory tests.
Postpartum hemorrhage | Within 24h after delivery
  Postpartum bleeding volume ≥500 mL.
Hepatic diseases | During pregnancy, delivery or within 42 days of pregnancy termination, an average of 1 year
  Hepatitis-B/C/E virus infection, acute fatty liver disease, or severe hepatitis.
Hematological diseases | During pregnancy, delivery or within 42 days of pregnancy termination, an average of 1 year
  Iron-deficiency anemia, thalassemia, hemophilia, idiopathic thrombocytopenic purpura, aplastic anemia, or disseminated intravascular coagulation.
Gynecological diseases | During pregnancy, delivery or within 42 days of pregnancy termination, an average of 1 year
  Uterine fibroids, ovarian cyst, cervical carcinoma, pelvic inflammation, or ovarian carcinoma.
Respiratory diseases | During pregnancy, delivery or within 42 days of pregnancy termination, an average of 1 year
  Pneumonia, bronchitis, asthma or pulmonary tuberculosis.
Thyroid disease | During pregnancy, delivery or within 42 days of pregnancy termination, an average of 1 year
  Hyperthyroidism or hypothyroidism.
ICU admission | During pregnancy, delivery or within 42 days of pregnancy termination, an average of 1 year
  Admission to intensive care unit.
Maternal death | During pregnancy, delivery or within 42 days of pregnancy termination, an average of 1 year
  Maternal death.
Macrosomia | within 1 month after delivery
  Birth weight >4000 g.
Infant of low-birth weight | within 1 month after delivery
  Birth weight <2500 g.
Neonatal ICU admission | Within 1 month after delivery
  Admission to neonatal intensive care unit.
Neonatal death | Within 1 month after delivery
  Neonatal death.
Large for gestational age | Within 1 month after delivery
  Neonatal weight, length, or head circumference above the 90th percentile for that gestational age.
Small for gestational age | Within 1 month after delivery
  Neonatal weight, length, or head circumference below the 10th percentile for that gestational age.
Neonatal defect | Within 1 month after delivery
  Neonatal defect.
Maternal adverse outcomes | During pregnancy, delivery or within 42 days of pregnancy termination, an average of 1 year
  There occurred one or more of preeclampsia, eclampsia, ICP, placenta previa, gestational diabetes, ruptured uterus, placental abruption, postpartum hemorrhage, hepatic diseases, hematological diseases, gynecological diseases, respiratory diseases, thyroid disease, ICU admission, or maternal death.
Neonatal adverse outcomes | Within 1 month after delivery
  There occurred one or more of macrosomia, low-birth weight, neonatal ICU admission, neonatal death, large for gestational age, small for gestational age, or neonatal defect.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, Doctor, Principal Investigator — Chinese Evidence-based Medicine Center, West China Hospital, Sichuan University

IPD SHARING:
Plan to Share IPD: Undecided